CLINICAL TRIAL: NCT00256607
Title: CSP #465A - Non-Traditional Cardiovascular Risk Factors And Atherosclerosis In Type 2 Diabetes
Brief Title: Non-traditional Cardiovascular Risk Factors and Atherosclerosis in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 465A
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary artery calcium (CAC): Cohort from the VADT study, had baseline coronary atherosclerosis assessed by coronary artery calcium (CAC) measured by computed tomography. Participants were followed over the 7.5-year study for development of cardiovascular endpoints.

SUMMARY:
A predominant consequence of diabetes mellitus (DM) type 2 is accelerated development of atherosclerosis related conditions. Conventional cardiovascular risk factors only explain a portion of the excess risk for atherosclerosis in this population. In vitro, animal and epidemiologic studies have suggested that a variety of "novel" cardiovascular risk factors (CVRF), including triglyceride-rich lipoproteins (TGRL), small dense low density lipoprotein (D-LDL) subfractions, oxidative stress, and advanced glycation endproduct (AGE) formation may contribute to the development of atherosclerosis. These risk factors may also induce endothelial cell activation/injury or local or systemic inflammation that cause elevations in plasma levels of additional novel risk factors, such as soluble adhesion molecules, plasminogen activator inhibitor-1 (PAI-1), fibrinogen and C-reactive protein (CRP). Many of these risk factors are increased in DM type 2, presumably as a consequence of hyperglycemia and insulin resistance. However, no studies have evaluated the singular or synergistic relationship of these novel (CVRF) to measures of atherosclerosis as well as to the development of clinical macrovascular events in individuals with diabetes. If, as we suspect, these novel CVRF are related to development of atherosclerosis and macrovascular disease, it will be critical for the future design of prevention strategies to know whether intensive glucose lowering significantly reduces the levels of these novel CVRF. Furthermore, it would be important to explore whether the relationship of the above novel risk factors to atherosclerosis and development of clinical events is attenuated in those individuals receiving glucose lowering therapy. Alternatively, if glucose lowering has no effect (or a negative effect), on relevant novel CVRF, this could potentially explain the limited success of intensive glucose lowering to reduce macrovascular events in several prior trials.

The investigator proposes to take advantage of the study population and framework of the recently approved VA Cooperative Study of "Glycemic Control and Complications in Diabetes Mellitus Type 2" to address these issues in an efficient and cost-effective manner.

DETAILED DESCRIPTION:
Primary Hypothesis:Hypothesis The novel CVRF including the selected indicators of artery wall injury and local or systemic inflammation, are related to the presence and development of atherosclerosis and macrovascular events in DM type 2.

2.Intensive glucose lowering therapy will reduce the levels of several, if not all, of the novel CVRF.

Secondary Hypotheses:

Primary Outcomes:

1. MYOCARDIAL INFARCTION: Myocardial infarctions (MI) will be determined based on the algorithm supplied at the end of this appendix. All suspected MI will be evaluated in detail by the Endpoints Committee. All supporting documentation, i.e., ECGs, hospital records, laboratory values, etc. needed to confirm or rule out the presence or absence of an MI will be obtained by personnel at the ECG Laboratory.
2. CONGESTIVE HEART FAILURE: Diagnosis of new congestive heart failure (CHF) can be made in the presence of at least two minor manifestations or new onset of pulmonary congestion requiring treatment. Treatment with diuretic, digitalis glycoside, ACE inhibitor, or hospitalization for management of symptoms of CHF would be appropriate.

Study Abstract:

Objectives A predominant consequence of diabetes mellitus (DM) type 2 is accelerated development of atherosclerosis related conditions. Conventional cardiovascular risk factors only explain a portion of the excess risk for atherosclerosis in this population. In vitro, animal and epidemiologic studies have suggested that a variety of "novel" cardiovascular risk factors (CVRF), including triglyceride-rich lipoproteins (TGRL), small dense low density lipoprotein (D-LDL) subfractions, oxidative stress, and advanced glycation endproduct (AGE) formation may contribute to the development of atherosclerosis. These risk factors may also induce endothelial cell activation/injury or local or systemic inflammation that cause elevations in plasma levels of additional novel risk factors, such as soluble adhesion molecules, plasminogen activator inhibitor-1 (PAI-1), fibrinogen and C-reactive protein (CRP). Many of these risk factors are increased in DM type 2, presumably as a consequence of hyperglycemia and insulin resistance. However, no studies have evaluated the singular or synergistic relationship of these novel (CVRF) to measures of atherosclerosis as well as to the development of clinical macrovascular events in individuals with diabetes. If, as we suspect, these novel CVRF are related to development of atherosclerosis and macrovascular disease, it will be critical for the future design of prevention strategies to know whether intensive glucose lowering significantly reduces the levels of these novel CVRF. Furthermore, it would be important to explore whether the relationship of the above novel risk factors to atherosclerosis and development of clinical events is attenuated in those individuals receiving glucose lowering therapy. Alternatively, if glucose lowering has no effect (or a negative effect), on relevant novel CVRF, this could potentially explain the limited success of intensive glucose lowering to reduce macrovascular events in several prior trials.

The investigator proposes to take advantage of the study population and framework of the recently approved VA Cooperative Study of "Glycemic Control and Complications in Diabetes Mellitus Type 2" to address these issues in an efficient and cost-effective manner.

Hypothesis

1. The above novel CVRF (outlined in Table 1), including the selected indicators of artery wall injury and local or systemic inflammation, are related to the presence and development of atherosclerosis and macrovascular events in DM type 2.
2. Intensive glucose lowering therapy will reduce the levels of several, if not all, of the novel CVRF.

Research Plan Specific objectives 1& 2: Cross-sectional observational objectives

1. Determine the cross-sectional relationship between baseline levels of novel CVRF and the presence of atherosclerosis as assessed by electron beam computed tomography measurement (EBCT) of coronary artery calcium (CAC) and abdominal aortic calcium (AAC).
2. Determine the cross-sectional relationship between baseline levels of novel CVRF and prevalence of clinical macrovascular disease.

Specific objective 3: Prospective interventional objective Determine whether intensive glucose lowering reduces levels of novel CVRF.

Future long-term specific objectives: Prospective observational objectives

1. Determine the ability of baseline levels, "on trial" levels, and change in levels of novel CVRF to predict progression of atherosclerosis.
2. Determine the ability of baseline levels, "on trial" levels, and change in levels of novel CVRF to predict clinical macrovascular events.

Results 89 cardiovascular events occurred during a median follow-up duration of 5.2 years. Although intensive glucose lowering therapy did not significantly reduce cardiovascular events in the substudy cohort as a whole, there was evidence that the response was modified by baseline CAC as indicated by significant p-values for treatment by log (CAC+1) interaction terms in unadjusted and multivariable adjusted models (0.01 and 0.03, respectively). Multivariable adjusted hazard ratios (HR) for the effect of treatment indicated a progressive diminution of benefit with increasing CAC. Subgroup analyses were also conducted for clinically relevant CAC categories, those above and below a Coronary Calcium score (Agatston score) of 100. For the subgroup with CAC > 100, 11 of 62 individuals had events, while only 1 of 52 individuals with CAC 100 suffered an event. The multivariable HR for intensive treatment for those with CAC > 100 was 0.74 (0.46-1.20, p=0.21), while for the subgroup with CAC 100, the corresponding HR was 0.08 (0.008- 0.77, p=0.03), with event rates of 39 and 4 per 1000 person-years, respectively.

Main Manuscript:Intensive Glucose Lowering Therapy Reduces Cardiovascular Disease Events in Veterans Affairs Diabetes Trial (VADT) Participants with Lower Calcified Coronary Atherosclerosis

ELIGIBILITY:
Inclusion Criteria:

- Patients with type 2 DM who are no longer responsive to maximum dose of one or more oral agents.

Exclusion Criteria:

* Patients that have not participated in the VADT.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study of patients who are enrolled in the ongoing randomized clinical trial AGlycemic Control and Complications in Diabetes Mellitus Type 2@
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
1) Determine the cross-sectional relationship between baseline levels of novel CVRF and the | 3 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Abraira, MD, Study Chair — Miami VA Healthcare System, Miami, FL
Locations (7):
- United States (7):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Medical Center, Long Beach, Long Beach, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Reaven PD, Moritz TE, Schwenke DC, Anderson RJ, Criqui M, Detrano R, Emanuele N, Kayshap M, Marks J, Mudaliar S, Harsha Rao R, Shah JH, Goldman S, Reda DJ, McCarren M, Abraira C, Duckworth W; Veterans Affairs Diabetes Trial. Intensive glucose-lowering therapy reduces cardiovascular disease events in veterans affairs diabetes trial participants with lower calcified coronary atherosclerosis. Diabetes. 2009 Nov;58(11):2642-8. doi: 10.2337/db09-0618. Epub 2009 Aug 3. PMID 19651816
- [Result] Reaven PD, Emanuele N, Moritz T, Klein R, Davis M, Glander K, Duckworth W, Abraira C; Veterans Affairs Diabetes Trial. Proliferative diabetic retinopathy in type 2 diabetes is related to coronary artery calcium in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2008 May;31(5):952-7. doi: 10.2337/dc07-1926. Epub 2008 Mar 3. PMID 18316393
- [Result] Reaven PD, Sacks J; Investigators for the VADT. Coronary artery and abdominal aortic calcification are associated with cardiovascular disease in type 2 diabetes. Diabetologia. 2005 Feb;48(2):379-85. doi: 10.1007/s00125-004-1640-z. Epub 2005 Feb 2. PMID 15688207
- [Result] Reaven PD, Sacks J; Investigators for the Veterans Affairs Cooperative Study of Glycemic Control and Complications in Diabetes Mellitus Type 2. Reduced coronary artery and abdominal aortic calcification in Hispanics with type 2 diabetes. Diabetes Care. 2004 May;27(5):1115-20. doi: 10.2337/diacare.27.5.1115. PMID 15111530
- [Result] Saremi A, Allison M, Ditomasso D, Ge L, Anderson R, Moritz TE, Duckworth W, Abraira C, Reaven PD; VADT. Preliminary report: hepatic fat and inflammation in type 2 diabetes mellitus. Metabolism. 2010 Mar;59(3):430-2. doi: 10.1016/j.metabol.2009.07.041. Epub 2009 Oct 21. PMID 19850309
- [Result] Saremi A, Moritz TE, Anderson RJ, Abraira C, Duckworth WC, Reaven PD; Veterans Affairs Diabetes Trial (VADT). Rates and determinants of coronary and abdominal aortic artery calcium progression in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2010 Dec;33(12):2642-7. doi: 10.2337/dc10-1388. Epub 2010 Aug 31. PMID 20807873
- [Result] Saremi A, Anderson RJ, Luo P, Moritz TE, Schwenke DC, Allison M, Reaven PD; VADT. Association between IL-6 and the extent of coronary atherosclerosis in the veterans affairs diabetes trial (VADT). Atherosclerosis. 2009 Apr;203(2):610-4. doi: 10.1016/j.atherosclerosis.2008.07.031. Epub 2008 Aug 5. PMID 18804762
- [Result] Saremi A, Bahn G, Reaven PD; VADT Investigators. Progression of vascular calcification is increased with statin use in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2012 Nov;35(11):2390-2. doi: 10.2337/dc12-0464. Epub 2012 Aug 8. PMID 22875226
- [Result] Koska J, Saremi A, Bahn G, Yamashita S, Reaven PD; Veterans Affairs Diabetes Trial Investigators. The effect of intensive glucose lowering on lipoprotein particle profiles and inflammatory markers in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2013 Aug;36(8):2408-14. doi: 10.2337/dc12-2082. Epub 2013 Mar 27. PMID 23536583